CLINICAL TRIAL: NCT02710175
Title: TSH and AMH in Infertile Women
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Haitham Hassan Ahmed, Maghagha general hospital, Ain Shams Maternity Hospital
Other Study IDs: HAhmed
Record Dates: First submitted 2015-12-30; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: serum TSH level

SUMMARY:
Infertility is defined as the inability of a couple to achieve pregnancy over an average period of one year (in women under 35 years of age) or 6 months (in women above 35 years of age) of unprotected sexual intercourse. Infertility can be due to female, male reasons or both. It can be either primary or secondary.

Thyroid dysfunction and autoimmune thyroiditis are known adverse risk factors for pregnancy as well as fertility, regardless of the presence of disease in women of reproductive age. In particular, hypothyroid women are at an increased risk of menstrual disorders and infertility because of altered peripheral estrogen metabolism, hyperprolactinaemia and abnormal release of gonadotropin-releasing hormone.

The prevalence of subclinical hypothyroidism characterized by aberrant high serum thyroid-stimulating hormone (TSH) levels with normal free thyroxin (FT4) levels in infertile women are reported to be approximately 20% and it is a primary cause of subfertility.

Indeed, average TSH levels in infertile women were reportedly higher than those in normal fertile women. And elevated serum TSH levels were associated with diminished ovarian reserve in infertile patients. Moreover, although levothyroxine replacement therapy for subclinical hypothyroidism in infertile patients remains debatable, thyroxin supplementation may improve fertility to successful pregnancy.

This data suggests that hypothyroidism is strongly correlated with infertility (Velkeniers et al., 2013).

On the other hand, female fecundity decreases with increasing age, primarily because of decreased ovarian function. Anti-mullerian hormone (AMH) is a dimeric glycoprotein belonging to the transforming growth factor-beta (TGF-B) super family, which act on tissue growth and differentiation. It is produced by the granulosa cells from pre-antral and small antral follicles. Ovarian research after oophorectomy showed that serum AMH levels were closely correlated with the number of primordial follicles; therefore, AMH is a suitable biomarker of ovarian age in women of reproductive age.

Expectedly, ovarian function may be affected by impaired thyroid function, although this association has not been elucidated. In this study, we will evaluate the relationship between thyroid function and AMH levels by comparing them in infertile patients and healthy fertile women.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-35 years
2. Diagnosed as primary infertility.
3. Duration of marriage more than 1 year.
4. Controls should be normal fertile women aged 20- 35 years had no history of treatment for infertility or thyroid disorders.

Exclusion Criteria:

1. Age: above 35 years old.
2. Women with ovarian dysfunction (PCO, post ovarian surgery).
3. Treated thyroid dysfunction (Autoimmune thyroiditis, hypothyroidism).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Ain shams maternity patients in infertility unit
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
TSH Levels in mIU/L | 1 year